CLINICAL TRIAL: NCT02939066
Title: Endoscopic Ultrasound-guided Needle-based Confocal Laser Endomicroscopy for Evaluation of Malignant Lymph Nodes - a Pilot Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Yanqing Li, Vice president of Qilu Hospital, Shandong University
Other Study IDs: 2016SDU-QILU-22
Record Dates: First submitted 2016-10-18; First posted 2016-10-19 (Estimated); Last update posted 2017-02-16 (Actual); Status verified 2017-02

CONDITIONS: Malignancy or Benign of Enlarged Lymph Nodes
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Current modalities for lymph node staging in cancer can be limited. Needle-based confocal laser endomicroscopy (nCLE) is a novel endoscopic technique, which is compatible with the 19-gauge FNA needle. Under endoscopic ultrasonography (EUS) guidance, nCLE enables real-time in vivo imaging of lesion tissues at cellular and subcellular levels.This study aimed to evaluate the feasibility of needle-based confocal laser endomicroscopy (nCLE) at the time of endoscopic ultrasound (EUS) and to describe the nCLE features that distinguish between benign and malignant lymph nodes.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing EUS for staging of malignancy or assessment of enlarged lymph nodes

Exclusion Criteria:

* Patients aged <18 years or >80 years
* Known allergy to fluorescein dye
* Previous EUS-FNA performed within the past 3 months, and usualcontraindications to EUS-FNA
* Pregnancy or breastfeeding
* Inability to provide informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients undergoing EUS for staging of malignancy or assessment of enlarged lymph nodes will be recruited in this study at Qilu Hospital, Shandong University.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2016-05; Primary Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
The nCLE interpretation criteria for the characterization of malignant lymph nodes | 20 months

CONTACTS AND LOCATIONS:
Overall Officials: Yanqing Li, PhD. MD., Study Director — Department of Gastroenterology, Qilu Hospital, Shandong University
Locations (1):
- Department of Gastroenterology, Qilu Hospital, Shandong University, Jinan, Shandong, China